CLINICAL TRIAL: NCT00865345
Title: An Inpatient Evaluation of Six-Day Subcutaneous Glucose Sensor Performance
Acronym: 6-DayFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 218
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes
Keywords: blood sugar; glucose; sensor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MMT-7003 subcutaneous glucose sensor — All subjects will use the glucose sensor, randomized to participate in a 12-hour frequent (15-minute) blood glucose sampling period on one of six days of sensor wear. Blood samples will be analyzed using a laboratory standard (YSI) for comparison to the glucose sensor to evaluate accuracy.
  Other Names: Glucose sensor; Blood sugar sensor; glucose monitor; blood sugar monitor; MiniMed sensor

SUMMARY:
The purpose of this study is to assess the performance of the subcutaneous glucose sensor over an extended sensor life. The sensor is currently approved for 3 days of use and this study will examine sensor safety and accuracy when used for six days. This study will also test sensor safety and accuracy when inserted in an alternate body location (buttock area in addition to abdomen area). The study hypothesis is that the sensor performance will not greatly diminish when used for six days, or in an alternate insertion area.

DETAILED DESCRIPTION:
The Medtronic MiniMed Subcutaneous Glucose Sensor was originally approved by the FDA for commercialization as part of the Continuous Glucose Monitoring System (CGMS) on June 15, 1999 (PMA 980022). The Sensor is composed of a microelectrode with a thin coating of glucose oxidase beneath several layers of biocompatible membrane. This same sensor is used as part of the Guardian REAL-Time System, the latest advance in continuous glucose monitoring, which is based on the CGMS. Similar to the CGMS, the Guardian REAL-Time System has been developed for use in conjunction with a standard home blood glucose meter. The Guardian REAL-Time received regulatory approval from the FDA in 2006.

As currently used, the Subcutaneous Glucose Sensor is labeled for a maximum use duration of 72 hours, using only the abdomen area as an insertion site. Recent studies have shown that the useful sensor life could extend beyond three days, and it is reasonable to expect a significant percentage of sensors to last six days. It is the goal of this study to confirm sensor performance accuracy data from one of these recent studies. The sensor is also commonly worn in body areas other than the abdomen (such as the buttock). This study will also demonstrate sensor accuracy when used in an alternate site.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 through 75 inclusive
* Type 1 Diabetes Mellitus treated using either CSII (continuous subcutaneous insulin infusion) or MDI (multiple daily injections) for a minimum of 3 months
* Willingness to perform required study and data collection procedures and adhere to operating requirements of the Guardian REAL-Time and CGMS iPro Systems
* Willingness to perform at least 4 capillary blood glucose tests per day while wearing the Guardian REAL-Time and iPro Systems
* Willing to participate in a 12 hour frequent blood sampling session during the study
* Subject agrees to comply with the study protocol requirements
* Informed Consent, HIPAA Authorization, and California Experimental Subject Bill of Rights (if applicable) signed by the subject
* The Subject is willing to wear both the Guardian REAL-Time and CGMS iPro Systems for 6 days (~144 hours).

Exclusion Criteria:

* The Subject has a history of tape allergies that have not been resolved
* The Subject has any skin abnormality (e.g. psoriasis, rash, staphylococcus infection) that has not been resolved and would inhibit them from wearing the sensors
* Any additional condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent the Subject from completing the study
* Subject is currently participating in an investigational study (drug or device)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mastrototaro, PHD, Study Director — Medtronic Diabetes
Locations (3):
- United States (3):
  - AMCR Institute, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Rainier Clinical Research Center, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous Sensor Group: All subjects wore subcutaneous sensors
Period: Overall Study
Arm/Group | Subcutaneous Sensor Group
Started | 63
Completed | 61
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Sensor Group
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 59
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 38.7 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Glucose Sensor Accuracy When Compared to Laboratory Standard (YSI-Yellow Springs Instruments)
Description: The primary accuracy parameter (primary effectiveness endpoint) was the comparative readings of paired sensor and YSI glucose readings, measured on days 1 through 6. Accuracy is defined as within 20% agreement between YSI and paired sensor (within 20 mg/dL if YSI <80 mg/dL). Accuracy ranges from 0 - 100, with higher number suggests better accuracy.
Time Frame: Days one through six of sensor use
Population: 61 subjects of 63 enrolled subjects (a total of 4971 paired YSI and sensor readings) completed participation in the inpatient frequent blood sampling procedure.
Measure: Number (95% Confidence Interval); unit: paired YSI/sensor glucose values
Units Other Than Participants: paired YSI/sensor glucose values
Groups:
- All Completed Subjects: All subjects that completed the inpatient frequent sampling procedure.
Arm/Group | All Completed Subjects
Number analyzed (Participants) | 61
Number analyzed (paired YSI/sensor glucose values) | 4971
paired YSI/sensor glucose values | 75.45 [69.48 to 81.43]
Statistical Analysis 1: Comparison: All Completed Subjects; Test type: Superiority or Other; p < 0.05, ANCOVA; null model ANOVA is used to calculate 95% CI around accuracy rate. Intercept was fit in the abscence of other predictors; Intercept from ANCOVA model = 70, 95% CI 2-sided [60 to 100], Standard Error of Mean 2

2. Secondary Outcome: Device Related Moderate or Device Related Severe Adverse Events
Description: Device related moderate adverse event: low level of inconvenience or concern to the subject and may interfere with daily activities but is usually improved by simple therapeutic remedy Device related severe adverse event: interrupts a subject's daily activity and typically requires intervening treatment. Note: device related determination is made by the site that there is a reasonable possibility that the adverse event may have been caused by the device.
Time Frame: days one through six of sensor wear
Measure: Number; unit: events
Arm/Group | All Completed Subjects
Number analyzed (Participants) | 61
events | 0

ADVERSE EVENTS:
Arm/Group | Subcutaneous Sensor Group
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 1/63
OTHER ADVERSE EVENTS (reported when occurring in more than 1.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Sensor Group (N=63)
Broken hand (Injury, poisoning and procedural complications) | 1 (1) — The 1 adverse event reported was a broken hand (right hand, fourth and fifth metacarpal fractured) which occurred when the subject intentionally "punched a truck."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days